CLINICAL TRIAL: NCT04052945
Title: Efficacy, Safety and Underlying Mechanisms of Sphenopalatine Ganglion Acupuncture for Seasonal Allergic Rhinitis: a Randomized, Double-blind, Placebo Controlled Study
Brief Title: Efficacy, Safety and Underlying Mechanisms of Sphenopalatine Ganglion Acupuncture for Seasonal Allergic Rhinitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Luo Zhang, Vice president, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPA acupuncture for SAR
Record Dates: First submitted 2019-08-03; First posted 2019-08-12 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Acupuncture; sphenopalatine ganglion; seasonal allergic rhinitis; neuropeptides; inflammatory cytokines; neuro-immune interactions
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPA acupuncture (Active Comparator): active SPG acupuncture plus rescue medication (AA group)
  Interventions: Procedure: SPA acupuncture
- sham acupuncture (Sham Comparator): sham-SPG acupuncture plus rescue medication (SA group)
  Interventions: Procedure: sham acupuncture

INTERVENTIONS:
Procedure: SPA acupuncture — For patients in the AA group, acupuncture was performed at a selected point in the SPG by inserting the needle from the lower border of the zygomatic arch, posterior to the suture protuberance between the zygomatic process and temporal process. The needle was directed obliquely anteriorly, until nearly the whole needle was beneath the skin, and then rotated until the patient felt "de-qi" sensations .
  The patients in the AA group received four courses of active acupuncture(visit 1,2,3 and 4) within first two weeks, and then followed-up for a further 2 weeks (visit 5 and visit 6 ).
  Arms: SPA acupuncture
Procedure: sham acupuncture — For patients in the SA group, the needle was inserted at the same acupuncture point as for patients in the AA group, but to a depth of only 2-3cm and the procedure of rotating, twirling and thrusting the needle was repeated. During the acupuncture process, the acupuncturist sat on the side of the participant, where the patient could neither see the acupuncturist's face nor the length of the needle.
  The patients in the SA group received four courses of active acupuncture(visit 1,2,3 and 4) with first two weeks, and then followed-up for a further 2 weeks (visit 5 and visit 6).
  Arms: sham acupuncture

SUMMARY:
In recent years, a number of randomized controlled trials have confirmed the efficacy and safety of acupuncture in the treatment of allergic rhinitis (AR). Indeed, the latest American clinical guidelines recommended acupuncture treatment for AR patients who are interested in non-pharmacological treatment.

In conventional acupuncture treatment for AR, needles are inserted at specific acupoints in the body; with several studies demonstrating acupuncture of sphenopalatine ganglion (SPG) to improve nasal symptoms and quality of life in nasal inflammatory diseases.

The investigators hypothesize that, compared with sham acupuncture and rescue medication (RM), active SPG acupuncture combined with RM would lead to greater improvements in symptoms score and reduction in overall need for antihistamines. To test this hypothesis the investigators design a randomized, double blind, controlled trial to evaluate the efficacy of SPG acupuncture in pollen-induced seasonal AR patients and to explore the potential underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. history of physician-diagnosed SAR with at least 2 years of typical symptoms, and TNSS>=6 at v0.
2. positive skin prick test (SPT) and/or positive serum antigen specific IgE to local seasonal pollens (Giant Ragweed, Mugwort, Goosefoot, etc)

Exclusion Criteria:

1. oral steroids within 4 weeks prior to recruitment
2. nasal steroids and/or antihistamine 2 weeks prior to recruitment
3. perennial AR
4. any respiratory infection within the previous 4 weeks prior to recruitment
5. history of nasal polyps, asthma or autoimmune disorders
6. previously received acupuncture therapy for AR within 1 month prior to recruitment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-03-25 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline symptom scores at visit 4 | Symptom scores will be assessed at baseline (V0), visit 4( V4). V4 is within 15 minutes after the fourth acupuncture.
  Patients recorded nasal and ocular symptom severity during the trial. Four nasal symptoms (itching, sneezing, rhinorrhoea and nasal obstruction) and two ocular symptoms (ocular itch and watery eyes) were individually graded on a ten-point scale (0, no symptoms; 1-3, mild symptoms; 4-7, moderate symptoms; 8-10, severe symptoms). Our primary outcome is TNSS change from baseline at the end of four-acupuncture treatment at Visit 4 (15 minutes after the fourth acupuncture ). The investigator will compare the symptom scores between the active acupuncture group and the sham acupuncture group.

SECONDARY OUTCOMES:
Rescue medication score | RMS will be assessed at baseline (V0), and each visit. V1 to V4 is within two weeks. V5 is one week after the fourth acupuncture, and V6 is two weeks after the fourth acupuncture. There is no acupuncture during both V5 and V6
  when the symptoms were very severe and could not tolerated, the patients could use loratadine as rescue medication. The need for rescue medication was assessed as rescue medication score (RMS), analyzed as the weekly sum of daily use of Loratadine (10mg/d, equivalent to 1 point) or nasal corticosteroid spray (2 points)
SNOT-22 | SNOT-22 will be assessed at baseline (V0), and each visit. V1 to V4 is within two weeks. V5 is one week after the fourth acupuncture, and V6 is two weeks later. There is no acupuncture during both V5 and V6.
  SNOT-22 is assessed to evaluate the quality of life of the SAR patients.
nasal patency | NCV, NAR and MCA will be assessed at baseline (V0), and each visit. V1 to V4 is within two weeks. V5 is one week after the fourth acupuncture, and V6 is two weeks after the fourth acupuncture.
  Eccovision acoustic rhinometry (Hood Labs, Pembroke, USA) was used to measure the total nasal cavity volume (NCV) and minimum cross-sectional area (MCA). The ATMO 300 Rhinomanometer (ATMOS MedizinTechnikGmbH&Co., Feldkirch, Germany) was used to measure the nasal airway resistance (NAR) by anterior active rhinomanometry.
neuropeptides in nasal secretions | Nasal secretions can be obtained at each visit. V1 to V4 is within two weeks. V5 is one week later and V6 is two weeks later. There is no acupuncture during both V5 and V6.
  The levels of neuropeptides; including substance P, vasoactive intestinal peptide (VIP) , neuropeptide Y (NPY)) will be analysed using ELISA.
inflammatory cytokines in nasal secretions | Nasal secretions can be obtained at each visit. V1 to V4 is within two weeks. V5 is one week later and V6 is two weeks later. There is no acupuncture during both V5 and V6.
  The levels of inflammatory cytokines; including interferon-γ (IFN-γ), tumor necrosis factor-α(TNF-α), interleukin (IL)-5, IL-8, IL-17A, and eotaxin in the supernatants will be analyzed using the Luminex System.
adverse events | adverse events will be recorded at V1 to V4. V1, V2, V3, and V4 is within two weeks. V5 is one week after fourth treatment and V6 is two weeks later. There is no acupuncture during both V5 and V6.
  Any adverse event following acupuncture was assessed by physicians and patients. Patients were instructed to record any unexpected signs, symptoms, and feelings during the entire trial period. the pain score will be recorded during V1-V4.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Hongfei Lou, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi SM, Park JE, Li SS, Jung H, Zi M, Kim TH, Jung S, Kim A, Shin M, Sul JU, Hong Z, Jiping Z, Lee S, Liyun H, Kang K, Baoyan L. A multicenter, randomized, controlled trial testing the effects of acupuncture on allergic rhinitis. Allergy. 2013 Mar;68(3):365-74. doi: 10.1111/all.12053. Epub 2012 Dec 18. PMID 23253122
- [Background] Xue CC, Zhang AL, Zhang CS, DaCosta C, Story DF, Thien FC. Acupuncture for seasonal allergic rhinitis: a randomized controlled trial. Ann Allergy Asthma Immunol. 2015 Oct;115(4):317-324.e1. doi: 10.1016/j.anai.2015.05.017. Epub 2015 Jun 11. PMID 26073163
- [Background] Wang K, Chen L, Wang Y, Wang C, Zhang L. Sphenopalatine Ganglion Acupuncture Improves Nasal Ventilation and Modulates Autonomic Nervous Activity in Healthy Volunteers: A Randomized Controlled Study. Sci Rep. 2016 Jul 18;6:29947. doi: 10.1038/srep29947. PMID 27425415
- [Background] Brinkhaus B, Ortiz M, Witt CM, Roll S, Linde K, Pfab F, Niggemann B, Hummelsberger J, Treszl A, Ring J, Zuberbier T, Wegscheider K, Willich SN. Acupuncture in patients with seasonal allergic rhinitis: a randomized trial. Ann Intern Med. 2013 Feb 19;158(4):225-34. doi: 10.7326/0003-4819-158-4-201302190-00002. PMID 23420231